CLINICAL TRIAL: NCT01845532
Title: Analgesic Effect of Trigger Point Injection and EMLA for Shoulder Pain in Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2013-0101
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Myoma of Uterus
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TPI group (Experimental)
  Interventions: Drug: TPI
- ELMA group (Active Comparator)
  Interventions: Drug: EMLA cream
- None group (No Intervention)

INTERVENTIONS:
Drug: TPI — Trigger point injection with 25G needle on the shoulder before surgery(0.5% procaine, 0.25~0.5% lidocaine, 0.125% bupivacaine)
  Other Names: Trigger Point Injection
  Arms: TPI group
Drug: EMLA cream — EMLA cream with occluding dressing on the shoulder before surgery(5% of eutectic mixture with 2.5% lidocaine and 2.5% prilocaine)
  Arms: ELMA group

SUMMARY:
Laparoscopic operative procedures have revolutionized gynecological surgery. These have several advantages: a smaller and more cosmetic incision, reduced blood loss and shorter postoperative stay, which cuts down on hospital costs. However, postoperative pain continues to be one complication, which results in an unpleasant experience for the patient and at times causes a delayed discharge. Trigger point injection removes the pain developing point and block the pain signal. EMLA cream shows analgesic effect when being spread on the skin. An literature showed that patch of local anesthetics showed the effect of trigger point inject. The purpose of this study is to investigate the alleviation of shoulder pain, headache, abdominal pain, and back pain after trigger point injection or EMLA cream applying on shoulder in patients undergoing total laparoscopic hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I or II
* age 20~70
* patients undergoing total laparoscopic hysterectomy

Exclusion Criteria:

* history of shoulder surgery
* coagulopathy
* infection or trauma of shoulder
* general inflammation
* allergy to local anesthetics

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
postoperative shoulder pain | 3 hr after end of surgery
  Postoperative shoulder pain is measured using the VAS at 3 hr after end of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea